CLINICAL TRIAL: NCT04683965
Title: A Single Arm, Open Label, Exploratory Study of Pemetrexed and TAS-102 in Combination With Bevacizumab in Patients Who Have Progressed After Standard Second Line Therapy
Brief Title: Pemetrexed and TAS-102 in Combination With Bevacizumab in Refractory Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEEP-G 06
Record Dates: First submitted 2020-12-22; First posted 2020-12-24 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Pemetrexed; trifluridine tipiracil drug combination; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pemetrexed + TAS-102 + Bevacizumab (Experimental): Pemetrexed 500 mg/m2 d1+ TAS-102, capsule, 35mg/m2, bid,po, d1~5, d8~12 + Bevacizumab 5 mg/kg d1, d14; Repeated every 4 weeks
  Interventions: Drug: Pemetrexed; Drug: TAS-102; Drug: Bevacizumab

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed 500 mg/m2 d1
Drug: TAS-102 — TAS-102, capsule, 35mg/m2, bid,p.o, d1~5,d8~12
  Other Names: LONSURF
Drug: Bevacizumab — Bevacizumab 5 mg/kg d1,d14
  Other Names: Avastin

SUMMARY:
Limited agents are optional after standard first and second line treatment for mCRC. Only Regorafenib and Fruquintinib are approved in China. PFS of these targeted drugs are not very long. Pemetrexed has shown significant efficacy in advanced lung cancer regarding PFS and OS with controllable toxicity. TAS-102 has been used in colorectal cancer with promising outcomes. Bevacizumab is also an important monoclonal antibody which could make benefits in treated patients. This study is aimed to explore the efficacy, safety in advanced colorectal cancer failed to standard therapy in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of adenocarcinoma of the colon or rectum. All other histological types are excluded.
* Subjects with metastatic colorectal cancer(CRC) (Stage IV).
* Subjects must have failed at least two lines of prior treatment, which must include a fluoropyrimidine, oxaliplatin and irinotecan.
* Subjects have failed or refused third-line treatment with regorafenib or fruquintinib.
* Subjects treated with oxaliplatin in an adjuvant setting should have progressed during or within 6 months of completion of adjuvant therapy.
* Subjects who have withdrawn from standard treatment due to unacceptable toxicity and precluding retreatment with the same agent prior to progression of disease will also be allowed.
* Prior treatment with bevacizumab and/or cetuximab will be allowed, but the use of bevacizumab should be no more than one single line treatment.
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1.is necessary.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
* Life expectancy of at least 3 months.
* Adequate bone marrow, liver, cardiac and renal function as assessed by the laboratory required by protocol.
* Assigned informed consent.

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
* Participants of other clinical trial within 4 weeks.
* Diseases which will impact the absorption of TAS-102, eg. dysphagia, chronic diarrhea, bowl obstruction
* Hemorrhage events of ≥grade 3 within 4 weeks.
* Known central nervous system metastasis.
* Uncontrolled hypertension. (Systolic blood pressure 140 mmHg or diastolic pressure 90 mmHg despite optimal medical management). Unstable angina,congestive heart failure,Myocardial infarction, Cardiac arrhythmias requiring anti-arrhythmic therapy.
* Urine protein ≥++ and 24h urine protein more than 1.0g.
* Chronically green wound or bone fracture.
* Arterial or venous thrombotic or embolic events.
* Tumor invading important blood vessel with high risk of severe hemorrhage.
* Current active bleeding or any surgery taken within 2 months.
* Abnormal coagulation function.
* Thromboemboli events within 6 months.
* Immune diseases or organ transplantation history.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | From assignment of the first subject to 3 months later after the last participant is recruited.The last participant will be recruited before November 1,2021
  The percentage of subjects with total number of Complete Response (CR) + total number of Partial Response (PR)

SECONDARY OUTCOMES:
Progression-free Survival(PFS) | From assignment of the first subject to 3 months later after the last participant is recruited.The last participant will be recruited before November 1,2021
  PFS was defined as the time from assignment to disease progression radiological/clinical or death due to any cause, whichever occurs first. Subjects without progression or death at the time of analysis were censored at their last date of tumor evaluation.
Overall Survival (OS) | From assignment of the first subject until 40 death events observed, up to 2 years.
  OS is defined as the time from date of assignment to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Disease control rate (DCR) | From assignment of the first subject to 3 months later after the last participant is recruited.The last participant will be recruited before November 1,2021
  DCR is defined as the percentage of subjects whose best response was not Progressive Disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR) + total number of Partial Response (PR) + total number of Stable Disease (SD)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From assignment of the first subject to 3 months later after the last participant is recruited.The last participant will be recruited before November 1,2021
  adverse events will be assessed according to CTCAE v4.0, including hematological and non-hematological adverse events. Non-hematological adverse events will be collected by patients reported outcomes questionaire. The adverse events of interest include hypertension,hand-foot syndrome,proteinuria,hoarseness,rash,etc.The dose reduction and drug discontinuance due to adverse events will also be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu XY, Huang XE, You SX, Lu YY, Cao J, Liu J. Phase II study of pemetrexed as second or third line combined chemotherapy in patients with colorectal cancer. Asian Pac J Cancer Prev. 2013;14(3):2019-22. doi: 10.7314/apjcp.2013.14.3.2019. PMID 23679311
- [Background] Passardi A, Fanini F, Turci L, Foca F, Rosetti P, Ruscelli S, Casadei Gardini A, Valgiusti M, Dazzi C, Marangolo M. Prolonged Pemetrexed Infusion Plus Gemcitabine in Refractory Metastatic Colorectal Cancer: Preclinical Rationale and Phase II Study Results. Oncologist. 2017 Aug;22(8):886-e79. doi: 10.1634/theoncologist.2017-0206. Epub 2017 Jun 7. PMID 28592624
- [Background] Lim SW, Lee S, Lee J, Park SH, Park JO, Park YS, Lim HY, Kang WK, Kim ST. Pemetrexed Monotherapy as Salvage Treatment in Patients with Metastatic Colorectal Cancer Refractory to Standard Chemotherapy: A Phase II Single-arm Prospective Trial. J Cancer. 2018 Jul 30;9(16):2910-2915. doi: 10.7150/jca.24948. eCollection 2018. PMID 30123359
- [Background] Yu Z, Wang J, Cai X, Gao Z, Wang S, Gu Y. Analysis of pemetrexed-based chemotherapy in the treatment of advanced colorectal cancer. Ann Transl Med. 2020 Nov;8(21):1368. doi: 10.21037/atm-20-1095. PMID 33313113